CLINICAL TRIAL: NCT05966363
Title: Comparison of Cone Beam Irradiation Versus Multi-detector Scanner for Ear Imaging
Acronym: ICSI
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/738
Record Dates: First submitted 2023-06-30; First posted 2023-07-28 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Irradiation; Adverse Effect
Keywords: irradiation; TDM; Cone Beam; CT; CBCT

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CBCT: Patients receiving a Cone Beam of the rocks as part of a cochlear implant position check at Besançon University Hospital
  Interventions: Radiation: Nanodot
- CT: Patients receiving a CT scan of the rocks at Besançon University Hospital, all indications combined
  Interventions: Radiation: Nanodot

INTERVENTIONS:
Radiation: Nanodot — Radiation measurements using nanodots placed on the eyes, ears, neck and lower abdomen during an imaging examination.

SUMMARY:
The primary objective of this study is to compare the irradiation between Cone Beam and CT of the petrous bone.

The primary endpoint is the measurement of equivalent doses per organ of interest (eyes, ears, thyroid and external genitalia).

The investigators have set up a prospective monocentric study. The investigators will measure irradiation of these different organs using nanodots placed on the patient during imaging.

The results of these measurements will be compared between Cone Beam (performed in the Besançon University Hospital ENT department for cochlear implant position checks) and CT (all indications combined).

ELIGIBILITY:
Inclusion Criteria:

* Adult or child patients of any gender and any age, including the pediatric population, receiving a CT scan of the petrous bone performed at Besançon University Hospital and prescribed in the Besançon University Hospital ENT department, or receiving a CBCT as part of an intraoperative check of cochlear implant position.
* Women menopausal for at least 24 months, surgically sterilized, or, for women of childbearing age, using an effective contraceptive method (oral contraceptives, contraceptive injections, intra-uterine devices, double-barrier method, contraceptive patches).
* Subject's non-opposition to study participation
* Affiliation with a French social security scheme or beneficiary of such a scheme.

Exclusion criteria are :

* Legal incapacity or limited legal capacity
* Subject unlikely to cooperate with the study and/or poor cooperation anticipated by the investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients are recruited during a consultation in the ENT department, either as part of a pre-cochlear implant assessment, or as part of a prescription for a CT scan of the petrous bone by the Besançon University Hospital ENT department department to be carried out at Besançon University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2023-07-26 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2024-09-19 (Actual)

PRIMARY OUTCOMES:
CT and CBCT induced Irradiation in ear imaging in adults with adult protocol | 9 month
  To compare CT and CBCT induced irradiation in ear imaging in adults and children > 15 years of age who have benefited from an adult protocol.

SECONDARY OUTCOMES:
CT and CBCT induced Irradiation in ear imaging in children with Pediatric protocol | 9 month
  To compare CT and CBCT induced irradiation in ear imaging in children ≤ 15 years of age who have benefited from a pediatric protocol.
CT and CBCT induced Irradiation in ear imaging in adults with pediatric protocol | 9 month
  To compare CT and CBCT induced irradiation in ear imaging in adults and children > 15 years of age who have benefited from a pediatric protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No